CLINICAL TRIAL: NCT01426009
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Seven Arm, Four-Period Cross-over, Incomplete Block Design, 7-Day Dosing Study to Assess the Dose-Response, Safety, and Efficacy of EP-101 (SUN101) in Subjects With Moderate to Severe COPD
Brief Title: Study to Investigate the Dose Response, Safety and Efficacy of Nebulized EP-101(SUN101) in Patients With Chronic Obstructive Pulmonary Disease (COPD): GOLDEN-1 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP-101-03
Record Dates: First submitted 2011-08-29; First posted 2011-08-30 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- EP-101 via nebulizer (eFlow®) 25 ug (Experimental): EP-101 via nebulizer (eFlow®)
  Interventions: Drug: EP-101 via nebulizer (eFlow®) 25 ug
- Tiotropium bromide via (Spiriva® Handihaler®) (Active Comparator): Tiotropium bromide via (Spiriva® Handihaler®)
  Interventions: Drug: Tiotropium bromide via (Spiriva® Handihaler®)
- Ipratropium bromide Inhalation Solution (Active Comparator): Ipratropium bromide Inhalation Solution via Handihaler® DPI
  Interventions: Drug: Ipratropium bromide Inhalation Solution via Handihaler® DPI
- Placebo EP-101 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo EP-101
- EP-101 via nebulizer (eFlow®) 50 ug (Experimental): EP-101 via nebulizer (eFlow®)
  Interventions: Drug: EP-101 via nebulizer (eFlow®) 50 ug
- EP-101 via nebulizer (eFlow®) 100 ug (Experimental): EP-101 via nebulizer (eFlow®)
  Interventions: Drug: EP-101 via nebulizer (eFlow®) 100 ug
- EP-101 via nebulizer (eFlow®) 200 ug (Experimental): EP-101 via nebulizer (eFlow®)
  Interventions: Drug: EP-101 via nebulizer (eFlow®) 200 ug

INTERVENTIONS:
Drug: EP-101 via nebulizer (eFlow®) 25 ug — EP-101 (25 ug ) Dose 1 administered once daily for 7 days
  Other Names: SUN101
  Arms: EP-101 via nebulizer (eFlow®) 25 ug
Drug: EP-101 via nebulizer (eFlow®) 50 ug — EP-101 (50 ug ) administered once daily for 7 days
  Other Names: SUN101
  Arms: EP-101 via nebulizer (eFlow®) 50 ug
Drug: EP-101 via nebulizer (eFlow®) 100 ug — EP-101 (100ug) administered once daily for 7 days
  Other Names: SUN101
  Arms: EP-101 via nebulizer (eFlow®) 100 ug
Drug: Placebo EP-101 — Placebo EP-101 administered once daily for 7 days
  Other Names: Placebo
  Arms: Placebo EP-101
Drug: Tiotropium bromide via (Spiriva® Handihaler®) — Tiotropium 18 µg administered once daily for 7 days using Handihaler® DPI
  Other Names: Tiotropium bromide
  Arms: Tiotropium bromide via (Spiriva® Handihaler®)
Drug: Ipratropium bromide Inhalation Solution via Handihaler® DPI — Ipratropium 500 µg administered three times daily for 7 days using general purpose nebulizer
  Other Names: Ipratropium bromide
  Arms: Ipratropium bromide Inhalation Solution
Drug: EP-101 via nebulizer (eFlow®) 200 ug — EP-101 (200) ug administered once daily for 7 days
  Other Names: SUN101
  Arms: EP-101 via nebulizer (eFlow®) 200 ug

SUMMARY:
The purpose of this study is to determine steady-state efficacy and dose response profile and to assess safety and pharmacokinetic profile of nebulized EP-101(SUN101) after 7-day dosing using an investigational high efficiency nebulizer (eFlow®) compared with placebo and two active comparators in patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This is a phase 2, multicenter, randomized, double-blind, placebo-controlled, four-period, incomplete block design cross-over study using EP-101(SUN101) and open-label active controls (tiotropium bromide and ipratropium bromide). The study population will consist of subjects of 40-75 years of age with moderate to severe COPD. Approximately 133 subjects diagnosed with moderate to severe COPD will be enrolled in order to achieve minimum 105 subjects completing the study.

Following a run-in phase, each subject will be randomly assigned to one of 7 treatment sequences,(96 sequences when order of administration is considered), with each sequence comprised of four 7-day Treatment Periods. There will be a washout period of 7 days between each Treatment Period. Study visits will be conducted on Days 1 and 7 of each Treatment Period, with an overnight stay required in the clinic during these visits. A Final Study Visit will be conducted 7 days following the last study treatment.

During each Treatment Period, study treatments will be administered once daily (QD), except for ipratropium inhalation solution, which will be administered three times daily (TID). EP-101 (SUN101)active and placebo treatments will be administered using an investigational high-efficiency eFlow® nebulizer. Tiotropium bromide (Spiriva®) will be administered in an open-label manner via Handihaler® dry-powder inhaler (DPI). Ipratropium bromide inhalation solution will be administered in an open-label manner via general purpose nebulizer.

This study was previously posted by Elevation Pharmaceuticals, Inc. On September 5, 2012, Elevation was acquired by merger with Sunovion Pharmaceuticals Inc. ("Sunovion"), which resulted in Elevation becoming a direct wholly-owned subsidiary of Sunovion. In conjunction with this acquisition, the name of Elevation has been changed to Sunovion Respiratory Development Inc.

ELIGIBILITY:
Inclusion Criteria:

* 40-75 years of age
* Clinical diagnosis of moderate to severe COPD
* Current/ex-smokers with at least 10 pack-year smoking history
* Post-bronchodilator FEV1 ≥ 30% and ≤ 70% predicted normal values
* Post-bronchodilator FEV1/FVC ratio of ≤ 0.70
* Post-bronchodilator improvement in FEV1 ≥ 12% and ≤ 30%, and a minimum of 100 mL
* Willing and able to remain at the study site for at least 24 hours at each study visit
* Signed written informed consent

Exclusion Criteria:

* Current evidence or recent history of any clinically significant and unstable disease or abnormality (e.g., myocardial infarction, cardiac failure, uncontrolled hypertension, life-threatening arrhythmias, uncontrolled diabetes)
* Primary diagnosis of asthma
* History of malignancy within the past 5 years
* History of COPD exacerbation within 6 weeks of Screening
* Daily oxygen therapy > 10 hours per day
* Systemic steroids use within 6 weeks of Screening
* Respiratory tract infection within 6 weeks of Screening
* History of tuberculosis, bronchiectasis
* History of urinary retention or bladder neck obstruction type symptoms
* History of glaucoma
* Prolonged QTc interval (>460msec) or history of long QT syndrome
* Recent history of alcohol or drug abuse
* Females who are pregnant or breastfeeding, or if of child-bearing potential unwilling to practice acceptable birth control methods
* History of hypersensitivity or intolerance to aerosol medications
* Participation in another investigational drug study within 30 days of Screening

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Tutuncu, M.D., Ph.D., Study Director — Chief Medical Officer / Elevation Pharmaceuticals, Inc.
Locations (11):
- United States (10):
  - Elevation Investigational Site, Phoenix, Arizona
  - Elevation Investigational Site, Los Angeles, California
  - Elevation Investigational Site, DeLand, Florida
  - Elevation Investigational SIte, Madisonville, Kentucky
  - Elevation Investigational Site, North Dartmouth, Massachusetts
  - Elevation Investigational Site, Charlotte, North Carolina
  - Elevation Investigational Site, Raleigh, North Carolina
  - Elevation Investigational Site, Medford, Oregon
  - Elevation Investigational Site, Spartanburg, South Carolina
  - Elevation Investigational Site, Tacoma, Washington
- Elevation Investigational Site, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One randomized subject did not receive any study medication.
Groups:
- Total: total subjects which includes:EP-101 via nebulizer (eFlow®), Tiotropium bromide via (Spiriva® Handihaler®), Ipratropium bromide Inhalation Solution via Handihaler® DPI , and Placebo EP-101",
Period: Period 1-First Intervention (7 Days)
Arm/Group | Total
Started | 139
EP-101 Via Nebulizer | 23
EP-101 Via Nebulizer | 24
EP-101 Via Nebulizer | 22
EP-101 Via Nebulizer | 23
Ipratropium Bromide | 23
Placebo | 24
Completed | 137
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Personal Reasons | 1
Period: Washout 1
Arm/Group | Total
Started | 137
Completed | 135
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Personal Reasons | 1
Period: Period 2-Second Intervention (7 Days)
Arm/Group | Total
Started | 135
EP-101 Via Nebulizer | 22
EP-101 Via Nebulizer | 24
EP-101 Via Nebulizer | 24
EP-101 Via Nebulizer | 23
Ipratropium Bromide | 21
Placebo | 21
Completed | 130
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — personal reasons | 1
Period: Washout 2
Arm/Group | Total
Started | 130
Completed | 129
Not Completed | 1
Not completed — electrive surgery | 1
Period: Period 3-Third Intervention (7 Days)
Arm/Group | Total
Started | 129
EP-101 Via Nebulizer | 19
EP-101 Via Nebulizer | 23
EP-101 Via Nebulizer | 22
EP-101 Via Nebulizer | 20
Ipratropium Bromide | 23
Placebo | 22
Completed | 129
Not Completed | 0
Period: Washout 3
Arm/Group | Total
Started | 129
Completed | 128
Not Completed | 1
Not completed — personal reasons | 1
Period: Period 4-Fourth Intervention (7 Days)
Arm/Group | Total
Started | 128
EP-101 Via Nebulizer | 10
EP-101 Via Nebulizer | 7
EP-101 Via Nebulizer | 8
EP-101 Via Nebulizer | 9
Ipratropium Bromide | 8
Tiotropium Bromide | 76
Placebo | 10
Completed | 127
Not Completed | 1
Not completed — personal reasons | 1
Period: Washout 4
Arm/Group | Total
Started | 127
Completed | 126
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: modified Intent to Treat population for analysis set
Groups:
- Total Particiants: total of all participants in the study
Arm/Group | Total Particiants
Number analyzed (Participants) | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 88
  >=65 years | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 138
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 134
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120
  United Kingdom | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in 24 Post Dose Trough Forced Expiratory Volume in 1 Second (FEV1)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines. Trough FEV1 was defined as the mean of the spirometry values collected at 23 hours 30 minutes and 24 hours post dose for Day 1 and Day 7 within each Treatment Period. Baseline was calculated as the mean of the FEV1 values at 45 minutes and 15 minutes prior to the morning dose at Day 1 of each Treatment Period. Change from baseline was calculated as the trough FEV1 value minus the baseline for Day 1 and Day 7.
Time Frame: Day 1 and Day 7
Population: All subjects who received at least one dose of study medication and who had Day 1 pre-dose and Day 7 trough FEV1 values were included in the modified intent to treat analysis set
Measure: Mean (Standard Deviation); unit: liters
Groups:
- EP-101 Via Nebulizer (eFlow®) 25 mcg; EP-101 Via Nebulizer (eFlow®) 50 mcg; EP-101 Via Nebulizer (eFlow®)100 mcg; EP-101 Via Nebulizer (eFlow®) 200 mcg: EP-101 via nebulizer (eFlow®)
  EP-101 via nebulizer (eFlow®): EP-101 Dose 1 administered once daily for 7 days
  EP-101 via nebulizer (eFlow®): EP-101 administered once daily for 7 days
- Placebo: Placebo
  Placebo : Placebo administered once daily for 7 days
Arm/Group | EP-101 Via Nebulizer (eFlow®) 25 mcg | EP-101 Via Nebulizer (eFlow®) 50 mcg | EP-101 Via Nebulizer (eFlow®)100 mcg | EP-101 Via Nebulizer (eFlow®) 200 mcg | Ipratropium Bromide Inhalation Solution | Tiotropium Bromide Via (Spiriva® Handihaler®) | Placebo
Number analyzed (Participants) | 72 | 75 | 75 | 75 | 72 | 76 | 77
liters
  Trough FEV1 - day 1 | 0.0477 (0.16359) | 0.1009 (0.13261) | 0.0648 (0.14239) | 0.0632 (0.14965) | 0.0933 (0.18980) | 0.0740 (0.144441) | 0.0301 (0.14394)
  Trough FEV1 - day 7: number analyzed (Participants) | 72 | 75 | 73 | 72 | 72 | 76 | 77
  Trough FEV1 - day 7 | 0.0478 (0.18965) | 0.0699 (0.16909) | 0.0666 (0.15132) | 0.0840 (0.13842) | 0.0292 (0.16507) | 0.0564 (0.16356) | -0.155 (0.17934)
Statistical Analysis 1: Comparison: EP-101 Via Nebulizer (eFlow®) 25 mcg vs Placebo; An ANCOVA was used with change from baseline in trough FEV1 as the response,with factors for treatment, period, sequence, baseline as a covariate and a random effect for subject nested within sequence. A sample size of 30 subjects per comparison(133 total with dropouts)provides 90% power to detect a 0.12L difference in mean change trough FEV1 between active and placebo at an alpha of 0.05 using a 2-tailed t-test and assuming a within-subject standard deviation for change in trough FEV1 of 0.2; Test type: Superiority — Day 7 analysis; p = 0.0003, ANCOVA; Least Squares Mean Difference (SE) = 0.0723, 95% CI 2-sided [0.0347 to 0.1099], Standard Error of Mean 0.0188 — Standard Error of the Mean Difference
Statistical Analysis 2: Comparison: EP-101 Via Nebulizer (eFlow®) 50 mcg vs Placebo; An ANCOVA was used with change from baseline in trough FEV1 as the response,with factors for treatment, period, sequence, baseline as a covariate and a random effect for subject nested within sequence.A sample size of 30 subjects per comparison(133 total with dropouts)provides 90% power to detect a 0.12L difference in mean change trough FEV1 between active and placebo at an alpha of 0.05 using a 2-tailed t-test and assuming a within-subject standard deviation for change in trough FEV1 of 0.2; Test type: Superiority — Day 7 analysis; p = 0.0006, ANCOVA; Least Squares Mean Difference (SE) = 0.0676, 95% CI 2-sided [0.0307 to 0.1046], Standard Error of Mean 0.0184 — Standard Error of the Mean Difference
Statistical Analysis 3: Comparison: EP-101 Via Nebulizer (eFlow®)100 mcg vs Placebo; An ANCOVA was used with change from baseline in trough FEV1 as the response, with factors for treatment, period, sequence, baseline as a covariate and a random effect for subject nested within sequence.A sample size of 30 subjects per comparison(133 total with dropouts)provides 90% power to detect a 0.12L difference in mean change trough FEV1 between active and placebo at an alpha of 0.05 using a 2-tailed t-test and assuming a within-subject standard deviation for change in trough FEV1 of 0.2; Test type: Superiority — Day 7 analysis; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1021, 95% CI 2-sided [0.0644 to 0.1398], Standard Error of Mean 0.0188 — Standard Error of the Mean Difference
Statistical Analysis 4: Comparison: EP-101 Via Nebulizer (eFlow®) 200 mcg vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority — Day 7 analysis; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1299, 95% CI 2-sided [0.0918 to 00.1681], Standard Error of Mean 0.0190 — Standard Error of the Mean Difference
Statistical Analysis 5: Comparison: Ipratropium Bromide Inhalation Solution vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority — Day 7 analysis; p = 0.0200, Mantel Haenszel; Least Squares Mean Difference (SE) = 0.0446, 95% CI 2-sided [0.0073 to 0.0820], Standard Error of Mean 0.0186 — Standard Error of the Mean Difference
Statistical Analysis 6: Comparison: Tiotropium Bromide Via (Spiriva® Handihaler®) vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority — Day 7 analysis; p = 0.0060, ANCOVA; Least Squares Mean Difference (SE) = 0.0813, 95% CI 2-sided [0.0243 to 0.1382], Standard Error of Mean 0.0284 — Standard Error of the Mean Difference
Statistical Analysis 7: Comparison: EP-101 Via Nebulizer (eFlow®) 25 mcg vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority — Day 1 analysis; p = 0.0402, ANCOVA; Least Squares Mean Difference (SE) = 0.0385, 95% CI 2-sided [0.0018 to 0.0752], Standard Error of Mean 0.0183 — Standard Error of the Mean Difference
Statistical Analysis 8: Comparison: EP-101 Via Nebulizer (eFlow®) 50 mcg vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority — Day 1 analysis; p = 0.0003, ANCOVA; Least Squares Mean Difference (SE) = 0.0696, 95% CI 2-sided [0.0337 to 0.1055], Standard Error of Mean 0.0179 — Standard Error of the Mean Difference
Statistical Analysis 9: Comparison: EP-101 Via Nebulizer (eFlow®)100 mcg vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority — Day 1 analysis; p = 0.0074, ANCOVA; Least Squares Mean = 0.0501, 95% CI 2-sided [0.0140 to 0.0861], Standard Error of Mean 0.0180

2. Primary Outcome: Standardized Change in FEV1 Area Under the Curve (AUC) (0-12hr , 12-24hr, 0-24hr) on Day 1 and Day 7
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines. The standardized FEV1 AUC(0-12hr and 12-24hr) on Day 1 and Day 7 was calculated using the trapezoidal rule from the changes in FEV1 at Day 1 and Day 7, respectively, from the baseline value (the mean of the two FEV1 values at 45 minutes and 15 minutes prior to morning dose at Day 1 of the respective Treatment Periods) and dividing by the actual length of the time interval.
Time Frame: Day 1 and Day 7
Population: All subjects who received at least one dose of study medication and who had Day 1 pre-dose and Day 7 trough FEV1 values were included in the modified intent-to-treat (mITT) analysis set
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | EP-101 Via Nebulizer (eFlow®) 25 mcg | EP-101 Via Nebulizer (eFlow®) 50 mcg | EP-101 Via Nebulizer (eFlow®)100 mcg | EP-101 Via Nebulizer (eFlow®) 200 mcg | Ipratropium Bromide Inhalation Solution | Tiotropium Bromide Via (Spiriva® Handihaler®) | Placebo
Number analyzed (Participants) | 72 | 76 | 75 | 71 | 74 | 75 | 76
liters
  AUC 0-12 on Day 1 | 0.1001 (0.15704) | 0.1520 (0.13646) | 0.1414 (0.11045) | 0.1720 (0.12644) | 0.1990 (0.13740) | 0.1213 (0.12548) | 0.0130 (0.11486)
  AUC 12-24 on Day 1 | 0.0039 (0.17104) | 0.0681 (0.12835) | 0.0413 (0.14032) | 0.0645 (0.13275) | 0.0987 (0.16958) | 0.0499 (0.14532) | -0.0245 (0.12151)
  AUC 0-24 on Day 1 | 0.0525 (0.15495) | 0.1107 (0.12207) | 0.0919 (0.11554) | 0.1194 (0.11905) | 0.1496 (0.14425) | 0.0872 (0.12638) | -0.0073 (0.11377)
  AUC 0-12 on Day 7 | 0.1034 (0.19035) | 0.1411 (0.16343) | 0.1329 (0.13416) | 0.1438 (0.14833) | 0.1603 (0.16420) | 0.1256 (0.15197) | -0.0098 (0.15537)
  AUC 12-24 on Day 7 | 0.0112 (0.18136) | 0.0540 (0.16633) | 0.0278 (0.15187) | 0.0614 (0.13450) | 0.0357 (0.17382) | 0.0283 (0.15596) | 0.0698 (0.16584)
  AUC 0-24 on Day 7 | 0.0579 (0.17822) | 0.0980 (0.15651) | 0.0812 (0.13293) | 0.1030 (0.13162) | 0.1009 (0.15882) | 0.0776 (0.14702) | -0.0395 (0.15415)
Statistical Analysis 1: Comparison: EP-101 Via Nebulizer (eFlow®) 25 mcg vs Placebo; ACU 0-24 on Day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.0767, 95% CI 2-sided [0.0505 to 0.1028], Standard Error of Mean 0.0131 — standard error of the mean difference
Statistical Analysis 2: Comparison: EP-101 Via Nebulizer (eFlow®) 50 mcg vs Placebo; ACU 0-24 Day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1220, 95% CI 2-sided [0.0965 to 0.1475], Standard Error of Mean 0.0127 — standard error of the Mean difference
Statistical Analysis 3: Comparison: EP-101 Via Nebulizer (eFlow®)100 mcg vs Placebo; AUC 0-24 Day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1222, 95% CI 2-sided [0.0965 to 0.1479], Standard Error of Mean 0.0128 — standard error of the Mean difference
Statistical Analysis 4: Comparison: EP-101 Via Nebulizer (eFlow®) 200 mcg vs Placebo; AUC 0-24 day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1625, 95% CI 2-sided [0.1362 to 0.1888], Standard Error of Mean 0.0131 — standard error of the Mean difference
Statistical Analysis 5: Comparison: Ipratropium Bromide Inhalation Solution vs Placebo; AUC 0-24 day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1690, 95% CI 2-sided [0.1434 to 0.1946], Standard Error of Mean 0.0128 — standard error of the Mean difference
Statistical Analysis 6: Comparison: Tiotropium Bromide Via (Spiriva® Handihaler®) vs Placebo; AUC 0-24 day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1095, 95% CI 2-sided [0.0716 to 0.1473], Standard Error of Mean 0.0189 — standard error of the Mean difference
Statistical Analysis 7: Comparison: EP-101 Via Nebulizer (eFlow®) 25 mcg vs Placebo; AUC 0-24 on Day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1095, 95% CI 2-sided [0.0812 to 0.1379], Standard Error of Mean 0.0141 — standard error of the Mean difference
Statistical Analysis 8: Comparison: EP-101 Via Nebulizer (eFlow®) 50 mcg vs Placebo; AUC0-24 on Day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1271, 95% CI 2-sided [0.0993 to 0.1548], Standard Error of Mean 0.0139 — standard error of the Mean difference
Statistical Analysis 9: Comparison: EP-101 Via Nebulizer (eFlow®)100 mcg vs Placebo; AUC 0-24 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1450, 95% CI 2-sided [0.1169 to 0.1730], Standard Error of Mean 0.0140 — standard error of the Mean difference
Statistical Analysis 10: Comparison: EP-101 Via Nebulizer (eFlow®) 200 mcg vs Placebo; AUC 0-24 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1688, 95% CI 2-sided [0.1403 to 0.1972], Standard Error of Mean 0.0142 — standard error of the Mean difference
Statistical Analysis 11: Comparison: Ipratropium Bromide Inhalation Solution vs Placebo; AUC 0-24 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1396, 95% CI 2-sided [0.1117 to 0.1730], Standard Error of Mean 0.0139 — standard error of the Mean difference
Statistical Analysis 12: Comparison: Tiotropium Bromide Via (Spiriva® Handihaler®) vs Placebo; AUC 0-24 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1183, 95% CI 2-sided [0.0795 to 0.1972], Standard Error of Mean 0.0194 — standard error of the Mean difference
Statistical Analysis 13: Comparison: EP-101 Via Nebulizer (eFlow®) 25 mcg vs Placebo; AUC 0-12 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1038, 95% CI 2-sided [0.0776 to 0.1301], Standard Error of Mean 0.0131 — standard error of the Mean difference
Statistical Analysis 14: Comparison: EP-101 Via Nebulizer (eFlow®) 50 mcg vs Placebo; AUC 0-12 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1468, 95% CI 2-sided [0.1212 to 0.1724], Standard Error of Mean 0.0128 — standard error of the Mean difference
Statistical Analysis 15: Comparison: EP-101 Via Nebulizer (eFlow®)100 mcg vs Placebo; AUC 0-12 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1579, 95% CI 2-sided [0.1322 to 0.1837], Standard Error of Mean 0.0128 — standard error of the Mean difference
Statistical Analysis 16: Comparison: EP-101 Via Nebulizer (eFlow®) 200 mcg vs Placebo; AUC 0-12 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1919, 95% CI 2-sided [0.1655 to 0.2184], Standard Error of Mean 0.0132 — standard error of the Mean difference
Statistical Analysis 17: Comparison: Ipratropium Bromide Inhalation Solution vs Placebo; AUC 0-12 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1994, 95% CI 2-sided [0.1738 to 0.2251], Standard Error of Mean 0.0128 — standard error of the Mean difference
Statistical Analysis 18: Comparison: Tiotropium Bromide Via (Spiriva® Handihaler®) vs Placebo; AUC 0-12 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1248, 95% CI 2-sided [0.0872 to 0.1625], Standard Error of Mean 0.0188 — standard error of the Mean difference
Statistical Analysis 19: Comparison: EP-101 Via Nebulizer (eFlow®) 25 mcg vs Placebo; AUC 0-12 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; standard error of the Mean difference; Least Squares Mean Difference (SE) = 0.1279, 95% CI 2-sided [0.0970 to 0.1587], Standard Error of Mean 0.0154 — standard error of the Mean difference
Statistical Analysis 20: Comparison: EP-101 Via Nebulizer (eFlow®) 50 mcg vs Placebo; AUC 0-12 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1454, 95% CI 2-sided [0.1151 to 0.1756], Standard Error of Mean 0.0151 — standard error of the Mean difference
Statistical Analysis 21: Comparison: EP-101 Via Nebulizer (eFlow®)100 mcg vs Placebo; AUC 0-12 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1699, 95% CI 2-sided [0.1393 to 0.2004], Standard Error of Mean 0.0152 — standard error of the Mean difference
Statistical Analysis 22: Comparison: EP-101 Via Nebulizer (eFlow®) 200 mcg vs Placebo; AUC 0-12 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1814, 95% CI 2-sided [0.1503 to 0.2125], Standard Error of Mean 0.0155 — standard error of the Mean difference
Statistical Analysis 23: Comparison: Ipratropium Bromide Inhalation Solution vs Placebo; AUC 0-12 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1697, 95% CI 2-sided [0.1393 to 0.201], Standard Error of Mean 0.0152 — standard error of the Mean difference
Statistical Analysis 24: Comparison: Tiotropium Bromide Via (Spiriva® Handihaler®) vs Placebo; AUC 0-12 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1384, 95% CI 2-sided [0.0951 to 0.1817], Standard Error of Mean 0.0216 — standard error of the Mean difference
Statistical Analysis 25: Comparison: EP-101 Via Nebulizer (eFlow®) 25 mcg vs Placebo; AUC 12-24 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.0471, 95% CI 2-sided [0.0155 to 0.0786], Standard Error of Mean 0.0157 — standard error of the Mean difference
Statistical Analysis 26: Comparison: EP-101 Via Nebulizer (eFlow®) 50 mcg vs Placebo; AUC 12-24 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.0918, 95% CI 2-sided [0.0611 to 0.1226], Standard Error of Mean 0.0154 — standard error of the Mean difference
Statistical Analysis 27: Comparison: EP-101 Via Nebulizer (eFlow®)100 mcg vs Placebo; AUC 12-24 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.0829, 95% CI 2-sided [0.0519 to 0.1139], Standard Error of Mean 0.0155 — standard error of the Mean difference
Statistical Analysis 28: Comparison: EP-101 Via Nebulizer (eFlow®) 200 mcg vs Placebo; AUC 12-24 o day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1299, 95% CI 2-sided [0.0982 to 0.1617], Standard Error of Mean 0.0158 — standard error of the Mean difference
Statistical Analysis 29: Comparison: Ipratropium Bromide Inhalation Solution vs Placebo; AUC 12-24 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1369, 95% CI 2-sided [0.1061 to 0.1678], Standard Error of Mean 0.0154 — standard error of the Mean difference
Statistical Analysis 30: Comparison: Tiotropium Bromide Via (Spiriva® Handihaler®) vs Placebo; AUC 12-24 on day 1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.0934, 95% CI 2-sided [0.0490 to 0.1377], Standard Error of Mean 0.0221 — standard error of the Mean difference
Statistical Analysis 31: Comparison: EP-101 Via Nebulizer (eFlow®) 25 mcg vs Placebo; AUC 12-24 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.0879, 95% CI 2-sided [0.0573 to 0.1186], Standard Error of Mean 0.0153 — standard error of the Mean difference
Statistical Analysis 32: Comparison: EP-101 Via Nebulizer (eFlow®) 50 mcg vs Placebo; AUC 12-24 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1088, 95% CI 2-sided [0.0788 to 0.1388], Standard Error of Mean 0.0150 — standard error of the Mean difference
Statistical Analysis 33: Comparison: EP-101 Via Nebulizer (eFlow®)100 mcg vs Placebo; AUC 12-24 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1175, 95% CI 2-sided [0.0872 to 0.1478], Standard Error of Mean 0.0151 — standard error of the Mean difference
Statistical Analysis 34: Comparison: EP-101 Via Nebulizer (eFlow®) 200 mcg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1532, 95% CI 2-sided [0.1226 to 0.1838], Standard Error of Mean 0.0153 — standard error of the Mean difference
Statistical Analysis 35: Comparison: Ipratropium Bromide Inhalation Solution vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.1048, 95% CI 2-sided [0.0747 to 0.1350], Standard Error of Mean 0.0150 — standard error of the Mean difference
Statistical Analysis 36: Comparison: Tiotropium Bromide Via (Spiriva® Handihaler®) vs Placebo; AUC 12-24 on day 7; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference (SE) = 0.0993, 95% CI 2-sided [0.0589 to 0.1398], Standard Error of Mean 0.0202 — standard error of the Mean difference

3. Secondary Outcome: Peak FEV1 (Maximum FEV1 During the First 4 Hours Post-dose on Day 1 and Day 7)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines
Time Frame: Day 1 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | EP-101 Via Nebulizer (eFlow®) 25 mcg | EP-101 Via Nebulizer (eFlow®) 50 mcg | EP-101 Via Nebulizer (eFlow®)100 mcg | EP-101 Via Nebulizer (eFlow®) 200 mcg | Ipratropium Bromide Inhalation Solution | Tiotropium Bromide Via (Spiriva® Handihaler®) | Placebo
Number analyzed (Participants) | 72 | 76 | 75 | 72 | 74 | 76 | 77
liters
  Day 1 | 1.469 (0.5049) | 1.498 (0.4857) | 1.443 (0.4431) | 1.455 (0.4355) | 1.601 (0.4665) | 1.434 (0.4774) | 1.356 (0.4471)
  Day 7 | 1.482 (0.4993) | 1.496 (0.4694) | 1.462 (0.4300) | 1.453 (0.4476) | 1.594 (0.4943) | 1.475 (0.4556) | 1.348 (0.4465)

4. Secondary Outcome: Treatment Responders (Number of Subjects With Clinically Meaningful Change From Pre-dose in Trough FEV1 on Day 1 and Day 7)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines. Clinically meaningful is defined as when the change from baseline (mean of the two pre-dose values at Day 1) in 24 hour trough FEV1 on a SUN-101 treatment is more than 100 mL compared to the mean change in trough FEV1 from all subjects on the placebo treatment.
Time Frame: Day 1 and Day 7
Population: All subjects who received at least one dose of study medication and who had Day 1 pre-dose and Day 7 through FEV1 values were included in the modified intent-to-treat (mITT) analysis set
Measure: Number; unit: number of participants
Arm/Group | EP-101 Via Nebulizer (eFlow®) 25 mcg | EP-101 Via Nebulizer (eFlow®) 50 mcg | EP-101 Via Nebulizer (eFlow®)100 mcg | EP-101 Via Nebulizer (eFlow®) 200 mcg | Ipratropium Bromide Inhalation Solution | Tiotropium Bromide Via (Spiriva® Handihaler®)
Number analyzed (Participants) | 72 | 76 | 75 | 72 | 74 | 76
number of participants
  Day 1 | 18 | 29 | 24 | 24 | 24 | 26
  Day 7 | 29 | 30 | 34 | 37 | 27 | 37

5. Secondary Outcome: Number of Participants With Adverse Events, Vital Signs, and Clinically Significant Abnormal ECG Values and Laboratory Tests
Description: AEs are defined as existing conditions which worsen or events which occur during the course of the clinical trial after treatment. Vital signs were performed during the screening period to confirm study eligibility and at the final study visit. ECGs were performed during the screening period to confirm study eligibility. Vital signs and ECG were additionally collected within 30 minutes pre-dose; and 30 minutes, and 1, 2, 4, 6, 12 hours, and 23 hours 45 minutes post-dose within each treatment period. Clinical laboratory assessments were conducted during the screening period, at each study visit during each treatment period, and at the final study visit.
Time Frame: Day 1 through Day 7
Population: All subjects who received at least one dose of study medication were included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | EP-101 Via Nebulizer (eFlow®) 25 mcg | EP-101 Via Nebulizer (eFlow®) 50 mcg | EP-101 Via Nebulizer (eFlow®)100 mcg | EP-101 Via Nebulizer (eFlow®) 200 mcg | Ipratropium Bromide Inhalation Solution | Tiotropium Bromide Via (Spiriva® Handihaler®) | Placebo
Number analyzed (Participants) | 74 | 78 | 76 | 75 | 75 | 76 | 77
Participants
  Treatment emergent AEs | 23 | 23 | 28 | 26 | 19 | 12 | 25
  Clinical signicant abnormal vital signs | 0 | 0 | 2 | 0 | 1 | 0 | 1
  Clinically significant abnormal ECG values Day 1 | 10 | 7 | 13 | 11 | 5 | 8 | 6
  Clinically significant abnormal ECG values Day 7 | 7 | 5 | 8 | 11 | 3 | 8 | 7
  Clinicall significant abnormal lab valuesday1-day7 | 1 | 0 | 2 | 2 | 1 | 0 | 3

6. Secondary Outcome: Rescue Medication Use
Description: Mean number of puffs of daily rescue medication
Time Frame: Day 1 through Day 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: average daily number of puffs
Arm/Group | EP-101 Via Nebulizer (eFlow®) 25 mcg | EP-101 Via Nebulizer (eFlow®) 50 mcg | EP-101 Via Nebulizer (eFlow®)100 mcg | EP-101 Via Nebulizer (eFlow®) 200 mcg | Ipratropium Bromide Inhalation Solution | Tiotropium Bromide Via (Spiriva® Handihaler®) | Placebo
Number analyzed (Participants) | 72 | 76 | 75 | 72 | 74 | 76 | 77
average daily number of puffs | 1.34 (2.72) | 1.11 (1.89) | 1.48 (2.43) | 1.29 (2.70) | 1.42 (2.91) | 1.33 (3.01) | 1.59 (2.16)

7. Secondary Outcome: Treatment Responders (Percentage of Subjects With Clinically Meaningful Change From Pre-dose in Trough FEV1 on Day 1 and Day 7)
Description: percentage of subjects with clinically meaningful change from pre-dose in trough FEV1 on Day 1 and Day 7 Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines.
Time Frame: Day 1 and Day 7
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | EP-101 Via Nebulizer (eFlow®) 25 mcg | EP-101 Via Nebulizer (eFlow®) 50 mcg | EP-101 Via Nebulizer (eFlow®)100 mcg | EP-101 Via Nebulizer (eFlow®) 200 mcg | Ipratropium Bromide Inhalation Solution | Tiotropium Bromide Via (Spiriva® Handihaler®)
Number analyzed (Participants) | 72 | 76 | 75 | 72 | 74 | 76
percentage of participants
  Day 1 | 25.0 | 38.7 | 32.0 | 35.3 | 33.8 | 34.7
  Day 7 | 40.3 | 40.0 | 46.6 | 51.4 | 37.5 | 48.7

ADVERSE EVENTS:
Time Frame: day 1 through day 7
Description: existing conditions which worsen or events which occur during the course of the clinical trial after treatment with randomized study drug has started
Arm/Group | EP-101 Via Nebulizer (eFlow®) 25 mcg | EP-101 Via Nebulizer (eFlow®) 50 mcg | EP-101 Via Nebulizer (eFlow®)100 mcg | EP-101 Via Nebulizer (eFlow®) 200 mcg | Ipratropium Bromide Inhalation Solution | Tiotropium Bromide Via (Spiriva® Handihaler®) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/78 | 0/76 | 0/75 | 0/75 | 0/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 8/74 | 13/78 | 14/76 | 13/75 | 5/75 | 2/76 | 16/77
Other Adverse Events (participants affected / at risk) | 0/74 | 0/78 | 0/76 | 0/75 | 0/75 | 0/76 | 0/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EP-101 Via Nebulizer (eFlow®) 25 mcg (N=74) | EP-101 Via Nebulizer (eFlow®) 50 mcg (N=78) | EP-101 Via Nebulizer (eFlow®)100 mcg (N=76) | EP-101 Via Nebulizer (eFlow®) 200 mcg (N=75) | Ipratropium Bromide Inhalation Solution (N=75) | Tiotropium Bromide Via (Spiriva® Handihaler®) (N=76) | Placebo (N=77)
headache (Nervous system disorders) | 3 (4) | 3 (5) | 5 (5) | 4 (7) | 0 (0) | 2 (3) | 7 (9)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 10 (13) | 9 (15) | 9 (14) | 5 (5) | 1 (1) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the study is part of a multi-center study. The first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.